CLINICAL TRIAL: NCT06870188
Title: Evaluation of the Clinical Success of Direct Restorations of Endodontically Treated Posterior Teeth in the Presence of Parafunction: A Pilot Study
Acronym: Fibre
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatma Yilmaz, Asistant professor doctor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Fiber-reinforced-comp-pilot; 23/152/02/3/4 (Other Grant/Funding Number: SCIENTIFIC RESEARCH PROJECTS COORDINATION UNIT OF MUĞLA SITKI KOÇMAN UNIVERSITY RECTORATE)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Bruxism; Endodontically Treated Molar; Composite Restoration; Fiber Reinforced Composite
Keywords: Fiber reinforced resin composite; composite restoration; endodontically treated teeth; bruxism
MeSH Terms: conditions — Bruxism; Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: The study included premolar and molar teeth with Class 1 and Class 2 cavity types and a remaining wall thickness of at least 3 mm, which had undergone endodontic treatment from volunteer participants. The teeth randomly assigned were restored into two groups: Group 1: fiber-reinforced composite restoration (FRCR), Group 2: composite restoration (CR). The restorations were evaluated at 6 and 12 months using the FDI criteria.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fiber-reinforced composite restoration (FRCR) (Experimental): After the cavity preparation, an adhesive was applied to the tooth, and a short fiber-reinforced flowable composite resin (EverX flow, GC) was used as the dentin replacement material. It was then covered with posterior composite resin (Gneal Posterior, GC).
  Interventions: Other: Composite Restoration; Other: Clinical evaluation
- Composite restoration (CR) (Experimental): After the cavity preparation, an adhesive was applied to the tooth, and only posterior composite resin material (Gneal Posterior, GC) was used for filling whole of the cavity
  Interventions: Other: Composite Restoration; Other: Clinical evaluation

INTERVENTIONS:
Other: Composite Restoration — The study included premolar or molar teeth with Class 1 and Class 2 cavity types and a remaining wall thickness of at least 3 mm, which had undergone endodontic treatment from volunteer participants. The teeth randomly assigned were divided into two groups: Group 1: fiber-reinforced composite restoration (FRCR), Group 2: composite restoration (CR). Direct composite restorations with or without fiber reinforced material were applied. The restorations were evaluated at 6 and 12 months using the FDI criteria.
Other: Clinical evaluation — The restorations were evaluated by two experienced and fully blinded observers according to the functional, esthetic, and biological criteria. The criteria were scored from 1 to 5 (sufficient/acceptable= score 1 to 3, insufficient/inacceptable but repair possible= score 4, and insufficient/inacceptable but repair not possible/reasonable= score 5). Scores of 4 and 5 were considered as failure in the restoration.

SUMMARY:
The aim of this prospective, randomized, parallel-group clinical study is to compare the 6- and 12-month clinical performances of direct composite restorations applied to endodontically treated posterior teeth with or without the use of fiber-reinforced composite material in individuals with parafunctional habits.

Bruxism is a repetitive jaw-muscle activity characterized by clenching and/or grinding of teeth. The possible outcomes of bruxism include wear and/or fractures in the teeth and restorations. Therefore, the choice of restorative methods and materials for restorations in bruxist individuals is of great importance. Direct adhesive restorations are the first treatment option for endodontically treated teeth with no excessive material loss and/or those that have lost vitality due to trauma. Over the past decade, the use of fiber-reinforced materials has been recommended to prevent catastrophic fractures. Fiber-reinforced materials have been developed and introduced to the market based on the idea that a restorative material that distributes or absorbs stress in high-stress areas will protect the underlying tooth structure.

Although there are numerous studies on the mechanical durability of restorative treatments for endodontically treated teeth in cases with parafunctional habits, there are limited clinical studies regarding the clinical performance of these methods.

The study included 32 premolar or molar teeth with Class 1 and Class 2 cavity types and a remaining wall thickness of at least 3 mm, which had undergone endodontic treatment from volunteer participants. The teeth randomly assigned were divided into two groups (n=16): Group 1: fiber-reinforced composite restoration (EverX flow, GC) (FRCR), Group 2: composite restoration (Gneal Posterior, GC) (CR). The restorations were evaluated at 6 and 12 months using the FDI criteria.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers aged 18 and above Cases where restoration was performed immediately after the completion of root canal treatment on posterior teeth Endodontically treated posterior teeth that required replacement of the old restoration due to secondary caries or fractures Cases without pulpal symptoms Posterior teeth classified as Class 1 and Class 2 according to cavity classification Teeth with a remaining wall thickness of at least 3 mm Presence of parafunction Teeth with a natural tooth in the opposing arch and adjacent teeth on both proximal sides

Exclusion Criteria:

* Individuals who are not volunteers
* Cases with ongoing pulpal symptoms
* Posterior teeth with cusp loss
* Teeth with root canal filling that is at least 2 mm shorter than the radiographic apex
* Individuals unable to attend periodic follow-up visits
* Individuals with a Gingival Index score greater than 1
* Severe periodontal disease
* Presence of systemic diseases
* Individuals with allergic reactions to any of the materials to be used
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-02-21 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
clinical success | 6 and 12 months-follow-up
  The restorations were evaluated by two experienced and fully blinded observers according to the functional, esthetic and biological criteria according to the FDI criteria. The criteria were scored from 1 to 5 (sufficient/acceptable= score 1 to 3, insufficient/inacceptable but repair possible= score 4, and insufficient/inacceptable but repair not possible/reasonable= score 5). Scores of 4 and 5 were considered as failure in the restoration.

CONTACTS AND LOCATIONS:
Locations (1):
- Muğla Sıtkı Koçman University, Menteşe, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Deliperi S, Bardwell DN. Reconstruction of nonvital teeth using direct fiber-reinforced composite resin: a pilot clinical study. J Adhes Dent. 2009 Feb;11(1):71-8. PMID 19343930
- [Background] Meyenberg K. The ideal restoration of endodontically treated teeth - structural and esthetic considerations: a review of the literature and clinical guidelines for the restorative clinician. Eur J Esthet Dent. 2013 Summer;8(2):238-68. PMID 23712344
- [Background] Frater M, Forster A, Kereszturi M, Braunitzer G, Nagy K. In vitro fracture resistance of molar teeth restored with a short fibre-reinforced composite material. J Dent. 2014 Sep;42(9):1143-50. doi: 10.1016/j.jdent.2014.05.004. Epub 2014 May 21. PMID 24859462
- [Background] Carvalho MA, Lazari PC, Gresnigt M, Del Bel Cury AA, Magne P. Current options concerning the endodontically-treated teeth restoration with the adhesive approach. Braz Oral Res. 2018 Oct 18;32(suppl 1):e74. doi: 10.1590/1807-3107bor-2018.vol32.0074. PMID 30365615
- [Derived] Yilmaz F, Ozturk Z, Demirbas A, Kursun S. Evaluation of the clinical success of direct restorations of endodontically treated posterior teeth in the presence of parafunction: a 12-month pilot study. Head Face Med. 2025 Oct 10;21(1):70. doi: 10.1186/s13005-025-00546-1. PMID 41068790